CLINICAL TRIAL: NCT01822574
Title: Effect of Surgical Technique on Resection Symmetry of the Patella in Total Knee Arthroplasty
Brief Title: Comparison of Three Surgical Techniques to Achieve Patella Symmetry During Resection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Robert T. Trousdale, MD, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-008219
Record Dates: First submitted 2013-03-18; First posted 2013-04-02 (Estimated); Results first posted 2016-03-02 (Estimated); Last update posted 2016-03-02 (Estimated); Status verified 2016-02

CONDITIONS: Arthroplasty, Replacement, Knee; Injuries, Knee
MeSH Terms: conditions — Knee Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cutting Guide Technique (Active Comparator): The guide is clamped onto the patella and tightened so that it remains stable. The guide has a slot that allows insertion of a standard sagittal saw blade, and this slot guides the blade as it is advanced across the patella. The thickness is then measured in the center of the patella to ensure that the resection goal is achieved. Additional resection may be performed as needed.
  Interventions: Procedure: Cutting Guide Technique
- Haptic Feedback Technique (Active Comparator): It consists of a free hand cut (no guide used) with a standard sagittal saw that is oriented based on osteo-cartilaginous landmarks and haptic palpation of the patella by the surgeon. The resection thickness/obliquity can be altered based on haptic feedback (use of the sense of touch) of the patella. The thickness is then measured in the center of the patella to ensure that the resection goal is achieved. Additional resection may be performed as needed.
  Interventions: Procedure: Haptic Feedback Technique
- Four Quadrant Technique (Active Comparator): Resection is performed in a free handed fashion, but after resection, the thickness of the patella is measured separately in all four quadrants (superolateral, superomedial, inferomedial, and inferolateral). Additional resection is performed as needed based on the quadrant measurements and the measurements are repeated after each resection until satisfactory resection thickness and symmetry are obtained.
  Interventions: Procedure: Four Quadrant Technique

INTERVENTIONS:
Procedure: Cutting Guide Technique — The guide is clamped onto the patella and tightened so that it remains stable. The guide has a slot that allows insertion of a standard sagittal saw blade, and this slot guides the blade as it is advanced across the patella. The thickness is then measured in the center of the patella to ensure that the resection goal is achieved. Additional resection may be performed as needed.
  Arms: Cutting Guide Technique
Procedure: Haptic Feedback Technique — It consists of a free hand cut (no guide used) with a standard sagittal saw that is oriented based on osteo-cartilaginous landmarks and haptic palpation of the patella by the surgeon. The resection thickness/obliquity can be altered based on haptic feedback (use of the sense of touch) of the patella. The thickness is then measured in the center of the patella to ensure that the resection goal is achieved. Additional resection may be performed as needed.
  Arms: Haptic Feedback Technique
Procedure: Four Quadrant Technique — Resection is performed in a free handed fashion, but after resection, the thickness of the patella is measured separately in all four quadrants (superolateral, superomedial, inferomedial, and inferolateral). Additional resection is performed as needed based on the quadrant measurements and the measurements are repeated after each resection until satisfactory resection thickness and symmetry are obtained.
  Arms: Four Quadrant Technique

SUMMARY:
This research was performed to determine which of the three techniques used by knee surgeons at the Mayo Clinic was the most accurate at the surgical removal (resection) of the knee-cap (patella) in a symmetric fashion during total knee replacement (arthroplasty). Although all three techniques are known to be effective, the three techniques had never been compared to one another to determine if one was more effective than the others at resecting the patella.

DETAILED DESCRIPTION:
Resection of the patella to prepare it for placement of a patellar prosthesis is a procedure that is performed routinely in the vast majority of total knee arthroplasties (TKA) in the United States and at the Mayo Clinic. This procedure is performed by a number of different techniques that have been proved to be safe and effective. Despite this, patellar instability, tilt, obliquity, and maltracking are all possible complications of improperly resected patellae during TKA. The goals of resection are to create a patella that is symmetrical, absent of obliquity (slanting), and thick enough to receive a patellar prosthesis. Although outcomes are generally good for most described methods, to date, little had been published regarding direct comparison of these methods.

Patients undergoing TKA with planned patellar resection were randomized to have their patella resected by one of three methods during primary TKA: 1) use of a cutting guide, 2) haptic feedback, or 3) free-hand resection guided by four quadrant measurements. There were three experienced fellowship-trained arthroplasty surgeons (hip and knee) performing the procedures who were all familiar and experienced with each of the three techniques being investigated. Each surgeon, within a group of 30 of their patients, performed a total 10 resections using each of the three methods listed above (30 resections per surgeon for a total of 90 resections).

Before and after resection measurements of knee-cap thickness were taken and used to determine patellar symmetry. The resulting symmetry of each of the three techniques was then be compared between and within each of the three techniques and surgeons. Each procedure was also be timed from first measurement by the staff surgeon to the final measurement by that surgeon.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for primary total knee arthroplasty with planned patellar resection by one of the three staff surgeons included in the study.
* Patient must be able and willing to provide consent for study participation

Exclusion Criteria:

* Patient in need of revision total knee arthroplasty or having already undergone prior total knee arthroplasty
* Patient not in need of patellar resection during their primary total knee arthroplasty
* Unwilling or unable to provide consent for participation

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2013-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Trousdale, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Camp CL, Martin JR, Krych AJ, Taunton MJ, Spencer-Gardner L, Trousdale RT. Resection Technique Does Affect Resection Symmetry and Thickness of the Patella During Total Knee Arthroplasty: A Prospective Randomized Trial. J Arthroplasty. 2015 Dec;30(12):2110-5. doi: 10.1016/j.arth.2015.05.038. Epub 2015 May 29. PMID 26115983

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the orthopedic department at Mayo Clinic in Rochester, Minnesota.
Period: Overall Study
Arm/Group | Cutting Guide Technique | Haptic Feedback Technique | Four Quadrant Technique
Started | 30 | 30 | 30
Completed | 30 | 30 | 30
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cutting Guide Technique | Haptic Feedback Technique | Four Quadrant Technique | Total
Number analyzed (Participants) | 30 | 30 | 30 | 90
Age, Continuous [Mean (Full Range); unit: years] | 71.1 [51.4 to 86.1] | 64.4 [42.0 to 72.2] | 67.3 [49.9 to 84.1] | 67.6 [42.0 to 86.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 14 | 18 | 48
  Male | 14 | 16 | 12 | 42
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 30 | 90

OUTCOME MEASURES:

1. Primary Outcome: Mean Asymmetry of the Patella After Patella Resection
Description: Post-resection symmetry of the patella was independently assessed by a resident or fellow who was not involved in the resection. This was evaluated by dividing the patella into four equal quadrants and measuring the thickness in the center of each quadrant using a ring tipped or "C"-shaped caliper. The difference between the thickest and thinnest measurements of the patella was reported as the value of asymmetry.
Time Frame: approximate average surgery time of 3 hours
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Cutting Guide Technique | Haptic Feedback Technique | Four Quadrant Technique
Number analyzed (Participants) | 30 | 30 | 30
mm | 1.73 (1.04) | 1.40 (0.88) | 0.85 (0.73)
Statistical Analysis 1: Comparison: Cutting Guide Technique vs Haptic Feedback Technique vs Four Quadrant Technique; A p-value less than 0.05 was considered statistically significant; Test type: Superiority or Other; p = 0.001, ANOVA

2. Secondary Outcome: The Difference Between Surgeon Goal and Actual Resection Height
Description: This outcome measure attempts to capture the most accurate method for obtaining a desired thickness. Each patellar resection procedure began by exposing the articular surface of the patella. Once the patella was fully exposed and the surgeon measured the native patellar thickness, the timer was started. The surgeon then stated their goal for post resection thickness, and these values were recorded. After the final resection, the timer was stopped. The ability to obtain the resection goal was independently assessed by a resident or fellow not involved in the resection. This was calculated by taking the difference between the surgeon's goal and the average thickness of the four quadrants measured by the resident or fellow.
Time Frame: Time 0 (prior to patella resection), and after surgery (approximately 3 hours)
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Cutting Guide Technique | Haptic Feedback Technique | Four Quadrant Technique
Number analyzed (Participants) | 30 | 30 | 30
mm | 1.40 (1.04) | 0.66 (0.64) | 0.66 (0.59)
Statistical Analysis 1: Comparison: Cutting Guide Technique vs Haptic Feedback Technique vs Four Quadrant Technique; A p-value less than 0.05 was considered statistically significant; Test type: Superiority or Other; p < 0.001, ANOVA

3. Secondary Outcome: Time to Complete Patella Resurfacing
Description: Each patellar resection procedure began by exposing the articular surface of the patella. Once the patella was fully exposed and the surgeon measured the native patellar thickness, the timer was started. After the final resection, the timer was stopped.
Time Frame: Time 0 (prior to patella resection), and after surgery (approximately 3 hours)
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Cutting Guide Technique | Haptic Feedback Technique | Four Quadrant Technique
Number analyzed (Participants) | 30 | 30 | 30
seconds | 128 (76.8) | 102 (34.7) | 110 (62.5)
Statistical Analysis 1: Comparison: Cutting Guide Technique vs Haptic Feedback Technique vs Four Quadrant Technique; A p-value less than 0.05 was considered statistically significant; Test type: Superiority or Other; p = 0.240, ANOVA

ADVERSE EVENTS:
Arm/Group | Cutting Guide Technique | Haptic Feedback Technique | Four Quadrant Technique
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes